CLINICAL TRIAL: NCT02378493
Title: Evaluation of the Antibiofilmogramme® Test During Diabetic Foot Infections
Acronym: BioFilm PieDia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: BioFilm Control (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: LOCAL/2014/AS-01b; 2014-A01745-42 (Other: ANSM)
Record Dates: First submitted 2015-02-23; First posted 2015-03-04 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Foot; Staphylococcus Aureus
Keywords: Antibiogramme; Antibiofilmogramme
MeSH Terms: conditions — Diabetic Foot; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure: Concordance between tests (Experimental): The study population is composed of diabetic patients with foot wounds (at least stage >=2) that are infected by at least 1 strain of S. aureus. Patients whose antibiogrammes and Antibiofilmogrammes are concordant will fall into this group (the "exposed" group).
  Upon inclusion, 1) all patients' wounds will be sampled, and 2) the associated bacterial strains identified via Vitek and 3) antibiograms performed; the latter are all part of routine procedure. 4) S. aureus isolates will be further analysed via an antiobiofilmogramme, which is an experimental element added by this research. At the end of the 1st regimen of antibiotics prescribed, if the treatment failed steps 1 to 4 can be repeated. 30 days after the end of the 1st regimen of antibiotics prescribed, steps 1 to 4 are systematically performed.
  Interventions: Biological: Antibiofilmogramme
- Non exposure: Not concordance between tests. (Experimental): The study population is composed of diabetic patients with foot wounds (at least stage >=2) that are infected by at least 1 strain of S. aureus. Patients who do not fall into the concordance (exposure) group, will fall into the non exposure group. The latter includes semi-concordance or discordance between antibiogrammes and Antiobiofilmogrammes.
  Upon inclusion, 1) all patients' wounds will be sampled, and 2) the associated bacterial strains identified via Vitek and 3) antibiograms performed; the latter are all part of routine procedure. 4) S. aureus isolates will be further analysed via an antiobiofilmogramme, which is an experimental element added by this research. At the end of the 1st regimen of antibiotics prescribed, if the treatment failed steps 1 to 4 can be repeated. 30 days after the end of the 1st regimen of antibiotics prescribed, steps 1 to 4 are systematically performed.
  Interventions: Biological: Antibiofilmogramme

INTERVENTIONS:
Biological: Antibiofilmogramme — An Antibiofilmogramme (BioFilm Control) evaluates the capacity of a series of antibiotics to inhibit the growth of bacterial biofilms for a given bacterial isolate.

SUMMARY:
This is an observational study that does not change routine care.

The primary objective of this study is to investigate the role of antibiogramme-antibiofilmogramme concordance (in terms of S. aureus strains and prescribed antibiotics) in the presence/absence of S. aureus strains at the end of a first regimen of antibiotics.

DETAILED DESCRIPTION:
The secondary objectives are:

A. Should a first regimen of antibiotics fail, to describe the bacterial community present in the wound, and its potential to create biofilms.

B. To investigate the role of antibiogramme-antibiofilmogramme concordance (in terms of S. aureus strains and prescribed antibiotics) in wound healing.

C. To study the potential role of additional antibiofilmogramme data, as well as that of other pre-defined co-factors, in predicting wound changes.

D. Create an S. aureus strain collection for future ancillary studies.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 7 to 10 weeks of follow-up
* Patient with a foot wound (at least stage 2 or more) that is infected by at least 1 strain of S. aureus

Exclusion Criteria:

* The patient is participating in, or has participated in within the past 3 months, another interventional study, or is currently in an exclusion period determined by a preceding study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Emergency situation precluding correct study implementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Presence/absence of S. aureus strains in the wound | At the end of 1st antibiotics (expected average of 21 days)
Antibiofilmogramme results | Baseline (Day 0)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance.
Antibiogram results | Baseline (Day 0)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance.

SECONDARY OUTCOMES:
Presence/absence of S. aureus strains in the wound | Baseline
Presence/absence of S. aureus strains in the wound | 30 days after end of 1st antibiotics (expected average of 51 days)
Antibiofilmogramme results | At the end of 1st antibiotics (expected average of 21 days)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance.
Antibiofilmogramme results | 30 days after end of 1st antibiotics (expected average of 51 days)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance.
Antibiogram results | At the end of 1st antibiotics (expected average of 21 days)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance.
Antibiogram results | 30 days after end of 1st antibiotics (expected average of 51 days)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance.
Wound surface area (mm^2) | Baseline (Day 0)
Wound surface area (mm^2) | At the end of 1st antibiotics (expected average of 21 days)
Wound surface area (mm^2) | 30 days after end of 1st antibiotics (expected average of 51 days)
Wound depth (mm) | Baseline (Day 0)
Wound depth (mm) | At the end of 1st antibiotics (expected average of 21 days)
Wound depth (mm) | 30 days after end of 1st antibiotics (expected average of 51 days)
The surface area of the wound has decreased by 40% compared to initial size: yes/no. | 30 days after end of 1st antibiotics (expected average of 51 days)
The number of bacterial strains detected in the wound. | Baseline (Day 0)
The number of bacterial strains detected in the wound. | At the end of 1st antibiotics (expected average of 21 days)
The number of bacterial strains detected in the wound. | 30 days after end of 1st antibiotics (expected average of 51 days)
The capacity of the S. aureus strains isolated to create biofilms in the presence of antibiotics | Baseline (Day 0)
  Score varying from 0 to 80
The capacity of the S. aureus strains isolated to create biofilms in the presence of antibiotics | At the end of 1st antibiotics (expected average of 21 days)
  Score varying from 0 to 80
The capacity of the S. aureus strains isolated to create biofilms in the presence of antibiotics | 30 days after end of 1st antibiotics (expected average of 51 days)
  Score varying from 0 to 80

OTHER OUTCOMES:
Age (years) | Baseline (Day 0)
Sex (m/f) | Baseline (Day 0)
Body mass index (kg/m^2) | Baseline (Day 0)
Antiobiotics taken | During the treatment period (expected average of 21 days)
% glycated hemoglobin | 30 days after end of 1st antibiotics (expected average of 51 days)
Systolic pressure index at the toe (ratio) | Baseline (Day 0)
Perception threshold for vibrations at the ankle (Hz) | Baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Sotto, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - CHU de Clermont-Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - CHU de Lyon - Hôpital de la Croix-Rousse, Lyon
  - CHU, Nantes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg

REFERENCES:
- [Result] Dunyach-Remy C, Ngba Essebe C, Sotto A, Lavigne JP. Staphylococcus aureus Toxins and Diabetic Foot Ulcers: Role in Pathogenesis and Interest in Diagnosis. Toxins (Basel). 2016 Jul 7;8(7):209. doi: 10.3390/toxins8070209. PMID 27399775